CLINICAL TRIAL: NCT04334967
Title: Randomized Study to Evaluate the Safety and Antiviral Efficacy of Hydroxychloroquine in Patients With Newly Diagnosed COVID-19 Compared to Standard of Care Treatment
Brief Title: Hydroxychloroquine in Patients With Newly Diagnosed COVID-19 Compared to Standard of Care
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: suspected unfavorable risk/benefit assessment
Sponsor: Providence Health & Services (Other)
Collaborators: Center for Outcomes Research and Education (Unknown); Providence Cancer Center, Earle A. Chiles Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020000186
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Corona Virus Infection; SARS-CoV-2; 2019-nCoV; 2019 Novel Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Hydroxychloroquine; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Upon confirmation of positive nasopharyngeal test for SARS-CoV-2, eligible patients will be randomized 1:1 to either a treatment group or control group.
Who Masked: Outcomes Assessor
Masking Description: Analysts will be blinded to patient randomization; outcome data analyses will be conducted with patient identifiers removed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Patients in the treatment arm will receive 200 mg oral hydroxychloroquine. Day 1: 400 mg doses twice (800 mg total). Days 2-5: 200 mg dose twice (400 mg total daily).
  Interventions: Drug: Hydroxychloroquine
- Control Arm (Active Comparator): Patients in the control arm will receive 500 mg oral Vitamin C. Day 1: 1000 mg dose twice (2000 mg total) Days 2-5: 500 mg dose twice (1000 mg total daily).
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Drug: Hydroxychloroquine — Treatment arm medication will be administered on an outpatient basis. Due to the emergent health crisis, study drug will be delivered to patients by institution staff or contract courier using a non-contact protocol.
  Arms: Treatment Arm
Dietary Supplement: Vitamin C — Control arm supplement will be administered on an outpatient basis. Due to the emergent health crisis, study supplies will be delivered to patients by institution staff or contract courier using a non-contact protocol.
  Other Names: ascorbic acid
  Arms: Control Arm

SUMMARY:
This study will assess the efficacy of hydroxychloroquine in reducing the severity of symptoms in patients with COVID-19

DETAILED DESCRIPTION:
Hydroxychloroquine has primarily been raised as a potential treatment of SARS-Cov-2 based on in vitro antiviral activity. A draft paper was released recently in March by Didier Raoult from Aix-Marseille University in France on a preliminary trial of 36 COVID-19 patients. In this trial, 6 patients were asymptomatic, 22 had upper respiratory symptoms, and 8 had lower respiratory symptoms. Between early and mid-March, they treated 20 of these patients with 600 mg of hydroxychloroquine daily in a hospital setting. Some patient also received the antibiotic azithromycin. 16 patients served as the controls. They observed a significant reduction in viral load in patients with hydroxychloroquine. After 6 days, 70% of the treated patients were considered cured (no virus detected in their samples) compared to 12.5% of controls. All 6 patients who received both hydroxychloroquine and azithromycin were negative for the virus after 6 days. This was an unblinded, non-randomized trial.

Vitamin C has multiple in-vivo effects on immune modulation that may, in sum, limit the development of the cytokine excess associated with critical illness. It is currently being studied in a clinical trial as a treatment for severe SARS-CoV-2 pneumonia in China and recommended as a supplement in standard treatment of COVID-19.

There are no medications currently approved for treatment of COVID-19. Hydroxychloroquine is a known drug with low toxicity that may reduce progression of respiratory symptoms and resulting hospitalizations. This randomized control study will assess its potential as an off-label treatment in reducing the rates of hospitalization and subsequent mechanical ventilation from COVID-19 infection compared to standard of care treatment with Vitamin C. A randomized control trial with placebo is impractical due to the increasing availability of this medication to the public.

ELIGIBILITY:
Inclusion Criteria:

* Must have positive nasopharyngeal swab for SARS-CoV-2 diagnosed via outpatient testing within the previous 48 hours
* Age ≥ 45 years
* Not hospitalized at the time of enrollment
* Established care with Providence provider
* Ability to understand a written or electronic informed consent document
* Reliable access to a computer or smartphone that can facilitate study communications via remote messaging or telephone and willingness to provide daily verbal check ins

Exclusion Criteria:

* Hypersensitivity to chloroquine or hydroxychloroquine
* History of retinal disease (macular degeneration, diabetic retinopathy, retinal rear/detachment, retinitis pigmentosa)
* History of seizure disorder
* History of ventricular tachycardia/fibrillation, history of long-QT syndrome, or ICD
* Current creatinine clearance <10 ml/min or on hemodialysis (as evidenced in EMR)
* Known G6PD deficiency
* Current use of the following medications: digoxin, amiodarone, flecainide, procainamide, oral dapsone. If other meds of concern, route to pharmacist to evaluate
* Concomitant use of the following only at Pharmacist/Investigator discretion: Abiraterone acetate, agalsidase, conivaptan, dabrafenib, dacomitinib, dapsone (systemic), digoxin, enzalutamide, fexinidazole, flecainide, fusidic acid (systemic), idelalisib, mifepristone, mitotane, pimozide, amiodarone, digoxin, procainamide, propafenone, stiripentol
* Currently on hospice
* Women of childbearing potential must not be pregnant, and must avoid becoming pregnant while on treatment and for 30 days following treatment discontinuation. Men must avoid fathering a child while on treatment and for 30 days following treatment discontinuation
* Any clinical factors such as bleeding, active infection, or psychiatric factors that in the judgment of the investigator would preclude safe participation and compliance with study procedures.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-05-27 (Estimated); Study Completion 2022-05-27 (Estimated)

PRIMARY OUTCOMES:
Total Hospitalization | 14 days
  This outcome will be assessed by comparing the percentages of enrolled patients that are hospitalized in the treatment and control arms.
Total Mechanical Ventilation | 14 days
  This outcome will be assessed by comparing the percentages of enrolled patients that have received mechanical ventilation in the treatment and control arms.

SECONDARY OUTCOMES:
Fever intensity measure | 2 days
  Self-reported body temperature. Each report scored low (less than 100.4), medium (100.4-102.2), or high (higher than 102.2). Outcome will be assessed by calculating percentage of patients with reported high, medium, low temperature at specified time points.
Fever intensity measure | 5 days
  Self-reported body temperature. Each report scored low (less than 100.4), medium (100.4-102.2), or high (higher than 102.2). Outcome will be assessed by calculating percentage of patients with reported high, medium, low temperature at specified time points.
Fever intensity measure | 10 days
  Self-reported body temperature. Each report scored low (less than 100.4), medium (100.4-102.2), or high (higher than 102.2). Outcome will be assessed by calculating percentage of patients with reported high, medium, low temperature at specified time points.
Fever intensity measure | 14 days
  Self-reported body temperature. Each report scored low (less than 100.4), medium (100.4-102.2), or high (higher than 102.2). Outcome will be assessed by calculating percentage of patients with reported high, medium, low temperature at specified time points.
Shortness of breath measure | 2 days
  Self-reported worsening shortness of breath. Each report scored yes/no. Outcome will be assessed by calculating percentage of patients with reported worsening of shortness of breath at specified time points.
Shortness of breath measure | 5 days
  Self-reported worsening shortness of breath. Each report scored yes/no. Outcome will be assessed by calculating percentage of patients with reported worsening of shortness of breath at specified time points.
Shortness of breath measure | 10 days
  Self-reported worsening shortness of breath. Each report scored yes/no. Outcome will be assessed by calculating percentage of patients with reported worsening of shortness of breath at specified time points.
Shortness of breath measure | 14 days
  Self-reported worsening shortness of breath. Each report scored yes/no. Outcome will be assessed by calculating percentage of patients with reported worsening of shortness of breath at specified time points.
Changes in daytime cough measure | 2 days
  Self reported changes in daytime cough. Each report scored 0 (no cough), 1 (one short coughing attack), 2 (two or more short coughing attacks), 3 (frequent coughing that did not interfere with activities), 4 (frequent coughing that did interfere with activities, 5 (distressing cough throughout most of the day). Outcome will be measured by calculating change in reported cough at each time point.
Changes in daytime cough measure | 5 days
  Self reported changes in daytime cough. Each report scored 0 (no cough), 1 (one short coughing attack), 2 (two or more short coughing attacks), 3 (frequent coughing that did not interfere with activities), 4 (frequent coughing that did interfere with activities, 5 (distressing cough throughout most of the day). Outcome will be measured by calculating change in reported cough at each time point.
Changes in daytime cough measure | 10 days
  Self reported changes in daytime cough. Each report scored 0 (no cough), 1 (one short coughing attack), 2 (two or more short coughing attacks), 3 (frequent coughing that did not interfere with activities), 4 (frequent coughing that did interfere with activities, 5 (distressing cough throughout most of the day). Outcome will be measured by calculating change in reported cough at each time point.
Changes in daytime cough measure | 14 days
  Self reported changes in daytime cough. Each report scored 0 (no cough), 1 (one short coughing attack), 2 (two or more short coughing attacks), 3 (frequent coughing that did not interfere with activities), 4 (frequent coughing that did interfere with activities, 5 (distressing cough throughout most of the day). Outcome will be measured by calculating change in reported cough at each time point.
Changes in nighttime cough measure | 2 days
  Self reported changes in nighttime cough. Each report scored 0 (no cough), 1 (cough on waking only), 2 (wake once or early due to cough), 3 (frequent waking due to cough), 4 (frequent coughing throughout the night, 5 (distressing cough preventing any sleep). Outcome will be measured by calculating change in reported cough at each time point.
Changes in nighttime cough measure | 5 days
  Self reported changes in nighttime cough. Each report scored 0 (no cough), 1 (cough on waking only), 2 (wake once or early due to cough), 3 (frequent waking due to cough), 4 (frequent coughing throughout the night, 5 (distressing cough preventing any sleep). Outcome will be measured by calculating change in reported cough at each time point.
Changes in nighttime cough measure | 10 days
  Self reported changes in nighttime cough. Each report scored 0 (no cough), 1 (cough on waking only), 2 (wake once or early due to cough), 3 (frequent waking due to cough), 4 (frequent coughing throughout the night, 5 (distressing cough preventing any sleep). Outcome will be measured by calculating change in reported cough at each time point.
Changes in nighttime cough measure | 14 days
  Self reported changes in nighttime cough. Each report scored 0 (no cough), 1 (cough on waking only), 2 (wake once or early due to cough), 3 (frequent waking due to cough), 4 (frequent coughing throughout the night, 5 (distressing cough preventing any sleep). Outcome will be measured by calculating change in reported cough at each time point.
Total mortality | 28 days
  Number of enrolled patients who have died within the specified time frame

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kendal, MD, Principal Investigator — Providence Medical Group Infectious Disease; Trista Johnson, PhD, MPH, Study Director — Providence Ambulatory Quality and Clinical Services
Locations (1):
- Portland Providence Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] CDC COVID-19 Response Team. Severe Outcomes Among Patients with Coronavirus Disease 2019 (COVID-19) - United States, February 12-March 16, 2020. MMWR Morb Mortal Wkly Rep. 2020 Mar 27;69(12):343-346. doi: 10.15585/mmwr.mm6912e2. PMID 32214079
- [Background] Cortegiani A, Ingoglia G, Ippolito M, Giarratano A, Einav S. A systematic review on the efficacy and safety of chloroquine for the treatment of COVID-19. J Crit Care. 2020 Jun;57:279-283. doi: 10.1016/j.jcrc.2020.03.005. Epub 2020 Mar 10. PMID 32173110
- [Background] Devaux CA, Rolain JM, Colson P, Raoult D. New insights on the antiviral effects of chloroquine against coronavirus: what to expect for COVID-19? Int J Antimicrob Agents. 2020 May;55(5):105938. doi: 10.1016/j.ijantimicag.2020.105938. Epub 2020 Mar 12. PMID 32171740
- [Background] Gao J, Tian Z, Yang X. Breakthrough: Chloroquine phosphate has shown apparent efficacy in treatment of COVID-19 associated pneumonia in clinical studies. Biosci Trends. 2020 Mar 16;14(1):72-73. doi: 10.5582/bst.2020.01047. Epub 2020 Feb 19. PMID 32074550
- [Background] Novel Coronavirus (2019-nCOV) Situation Report - 1. World Health Organization (WHO), 21 January 2020.
- [Background] Novel Coronavirus disease 2019 (2019-nCOV) Situation Report - 60. World Health Organization (WHO), 19 March 2020.
- [Background] Tricou V, Minh NN, Van TP, Lee SJ, Farrar J, Wills B, Tran HT, Simmons CP. A randomized controlled trial of chloroquine for the treatment of dengue in Vietnamese adults. PLoS Negl Trop Dis. 2010 Aug 10;4(8):e785. doi: 10.1371/journal.pntd.0000785. PMID 20706626
- [Background] Touret F, de Lamballerie X. Of chloroquine and COVID-19. Antiviral Res. 2020 May;177:104762. doi: 10.1016/j.antiviral.2020.104762. Epub 2020 Mar 5. PMID 32147496
- [Background] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618